CLINICAL TRIAL: NCT07278440
Title: ET-NEURO: A Pilot Trial of the Exercise Together Program in Primary Brain Tumor Patient-Caregiver Dyads Incorporating Glymphatic MRI
Brief Title: An Exercise Intervention for Improving Mental and Physical Health in Patients With Primary Brain Tumors and Their Caregivers, ET-NEURO Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Huan Vo, M.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00029300; NCI-2025-08714 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00029300 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2025-12-02; First posted 2025-12-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Primary Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy; Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (Exercise Together) (Experimental): Patients and caregivers participate in Exercise Together virtual resistance training sessions, over 75 minutes each, twice weekly for 12 weeks. Patients may undergo MRI throughout the study as part of their standard care.
  Interventions: Other: Electronic Health Record Review; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Other: Resistance Training

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Participate in Exercise Together
  Other Names: Strength Training

SUMMARY:
This clinical trial evaluates the effects of a partnered exercise program, called Exercise Together, on participants with primary brain tumors and their caregivers. Standard treatments for primary brain tumors require extensive caregiver support, and both patients and caregivers experience high psychological distress and physical burden as a result. While exercise is known to improve outcomes in cancer patients, its impact on primary brain tumor patients and caregivers remains unstudied. Exercise Together is a supervised, group exercise program previously studied in patients with other types of cancer, though never in patients with primary brain tumors or their caregivers. Exercise Together uses functional resistance training to target muscle groups essential for everyday activities to improve daily functioning. Since exercises are done in a partnered format, Exercise Together is also designed to foster teamwork and strengthen the relationship between the patient and their caregiver. This program may be safe, feasible, and effective in improving the mental and physical health of primary brain tumor patients and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and feasibility of the Exercise Together program for patient-participants with a diagnosis of primary brain tumor and their caregiver-participants.

SECONDARY OBJECTIVE:

I. To preliminarily evaluate the impact of the Exercise Together program on enhancing patient-caregiver relationships and improving quality of life in dyads affected with primary brain tumor (PBT).

EXPLORATORY OBJECTIVE:

I. To investigate the changes in the central nervous system (CNS) glymphatic system before, during, and after the exercise program and its association with cognition.

OUTLINE:

Patients and caregivers participate in Exercise Together virtual resistance training sessions, over 75 minutes each, twice weekly for 12 weeks. Patients may undergo magnetic resonance imaging (MRI) throughout the study as part of their standard care.

After completion of study intervention, participants are followed up at 4 weeks and then monthly in months 1-4.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT INCLUSION:
* Patient participants must have a histologically confirmed diagnosis of World Health Organization (WHO) grade 1-4 PBT such as glioblastoma, astrocytoma, oligodendroglioma, ependymoma, medulloblastoma, meningioma, and other primary brain tumors. Confirmed by review of the electronic medical record (EMR) and subsequently recorded in health history questionnaire. In cases where the EMR isn't clear, their Oregon Health & Science University OHSU provider will be contacted for confirmation
* Patient participants on active oral chemotherapy, including cytotoxic chemotherapy and molecularly targeted therapy, for the treatment of PBT are allowed
* Patient participants must be at least 6 weeks after the last dose of intravenous infusion chemotherapy for the treatment of PBT, including bevacizumab, prior to enrollment
* Patient participants must be at least 6 weeks post-radiation for PBT prior to enrollment. Patient participants must be at least 8 weeks post-craniotomy prior to enrollment
* Patient participants must have a co-residing spouse or partner caregiver due to the program's focus on intimacy
* Patient participants must have a Karnofsky performance score of at least 70 or an Eastern Cooperative Oncology Group (ECOG) score of 1 or less
* Patient participants are permitted to participate in other therapeutic interventional clinical trials for PBT
* PATIENT AND CAREGIVER INCLUSION:
* Patient participants and caregiver participants must be 18 years of age or older
* Patient participants and caregiver participants must state willingness to comply with all study procedures and availability for the duration of the study
* Patient participants and caregiver participants must have the ability to understand and the willingness to sign a written informed consent document
* Patient participants and caregiver participants must have home internet sufficient for videoconferencing

Exclusion Criteria:

* PATIENT AND CAREGIVER EXCLUSION:
* Patient and caregiver participants must not have engaged in two or more regular strength training sessions per week (e.g., physical therapy) during the past 30 days, as confirmed by self-report on the health history questionnaire
* Patient participants and caregiver participants with cognitive difficulties preclude answering survey questions. In the event of a suspected undeclared cognitive impairment, it will be confirmed by physician clearance or professional opinion of the principal investigator
* Patient participants and caregiver participants with medical condition, movement condition, pre-existing focal neurological deficits, new focal deficits concerning for recurrent or progressive PBT necessitating second line treatment, post operative deficits/wound, or medication use that contraindicates participation in moderate intensity exercise. Specific contraindications include the following: poorly controlled diabetes, recent cardiac event, neuromuscular disease, untreated orthostatic hypertension, recent surgery, acute hernia, acute rheumatoid arthritis, severe memory disorders, severe balance disorder, inability to ambulate without a walker or wheelchair, inability to stand for 3 minutes, severe hearing or vision problem

  * Confirmed by a combination of reviewing the EMR, self-report on the health history questionnaire, and/or by physician clearance. All patient participants will receive physician clearance by the neuro-oncology investigators prior to participating in the trial. For caregiver participants: must answer 'No' to American College of Sports Medicine pre-participation screening questions. If caregiver participants answer 'Yes' to either question they may be required to obtain physician clearance prior to being considered eligible. Physician clearance may also be requested at the discretion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate (feasibility) | Following screening at baseline
  Feasibility will be evaluated using an enrollment rate of ≥ 50% of eligible patient-caregiver dyads. Continuous variables will be characterized by N, mean or median, standard deviation or interquartile range; and discrete variables will be characterized by frequencies and proportions with exact 95% confidence intervals, as appropriate.
Adherence (feasibility) | Up to 12 weeks
  Feasibility will be evaluated using adherence, which will be defined as ≥ 50% of enrolled dyads completing at least 50% of the prescribed sessions (i.e., both members of the dyads attend ≥ 12 of 24 supervised exercise sessions). Continuous variables will be characterized by N, mean or median, standard deviation or interquartile range; and discrete variables will be characterized by frequencies and proportions with exact 95% confidence intervals, as appropriate.
Retention (feasibility) | Up to 4 weeks after intervention completion
  Feasibility will be evaluated using a retention rate of ≥ 50%. Continuous variables will be characterized by N, mean or median, standard deviation or interquartile range; and discrete variables will be characterized by frequencies and proportions with exact 95% confidence intervals, as appropriate.
Incidence of adverse events | Up to 1-month post-exercise intervention
  Defined as grade 3 or higher adverse events in both patient-participants and caregiver-participants, as per Common Terminology Criteria for Adverse Events version 5.0, directly attributable to the study intervention during the Exercise Together program. Continuous variables will be characterized by N, mean or median, standard deviation or interquartile range; and discrete variables will be characterized by frequencies and proportions with exact 95% confidence intervals, as appropriate.

SECONDARY OUTCOMES:
Quality of life | At baseline, 6 weeks, 12 weeks, and 16 weeks
  Appropriate summary statistics (e.g., mean or median, standard deviation or interquartile range) will be used to characterize quality of life measures at each time point for the following questionnaires for patient participants: Distress Thermometer (DT), Functional Assessment of Chronic Illness Therapy fatigue questionnaire, European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 together with the brain tumor-specific module. For caregiver participants, will use the following: DT, Short Form-36 questionnaire physical functioning subscale, as well as Caregiver Quality of Life Index-Cancer scale. Continuous variables will be characterized by N, mean or median, standard deviation or interquartile range; and discrete variables will be characterized by frequencies and proportions with exact 95% confidence intervals, as appropriate.
Patient and caregiver relationship quality | At baseline, 6 weeks, 12 weeks, and 16 weeks
  Will be measured using the dyadic coping measure. A linear mixed model will be used to quantify the trend over time and estimate the changes from baseline to each follow up time point. Hypothesis tests may be conducted for exploratory purposes and signal detection. Variation of time trend by patient characteristics may also be explored cautiously. Model assumptions will be checked and if not satisfied, alternative methods will be used. Continuous variables will be characterized by N, mean or median, standard deviation or interquartile range; and discrete variables will be characterized by frequencies and proportions with exact 95% confidence intervals, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Anh Huan Vo, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States